CLINICAL TRIAL: NCT01591148
Title: A High Resolution Pharmacokinetic/Pharmacodynamic Model of Propofol in Morbidly Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jerry Ingrande, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Stanford-16509; 16509-JI (Other: Stanford University)
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Morbid Obesity
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Obesity, Morbid | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morbidly obese subjects (Experimental): Morbidly obese subjects (body mass index greater than 40) will be given propofol for induction of general anesthesia. Plasma samples will be taken to ascertain drug concentration over time.
  Interventions: Drug: propofol
- Control subjects (body mass index 20-25) (Active Comparator): Normal weight subjects (body mass index 20-25) will be given propofol during induction of general anesthesia. Plasma samples will be collected over time to ascertain propofol plasma concentration.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Morbidly obese subjects (body mass index greater than 40)and control subjects (body mass index 20-25) will be given propofol for induction of general anesthesia. Plasma samples will be taken to ascertain drug concentration over time.

SUMMARY:
This study will determine how morbid obesity affects the distribution and metabolism of the drug propofol. The investigators hypothesize that propofol will be distributed and metabolized differently in morbidly obese subjects as compared to normal weight subjects.

ELIGIBILITY:
Inclusion Criteria:

* adult age (ages 18-70)
* body mass index greater than 40 or between 20-25
* American Society of Anesthesiologists Class I, II, or III
* undergoing elective surgical procedure requiring general anesthesia

Exclusion Criteria:

* evidence of cardiovascular or pulmonary disease
* kidney or liver dysfunction
* drug allergy to propofol
* history of difficult airway
* on prescribed or over the counter anxiolytics, antipsychotics, or sleeping aids
* unable to speak or understand English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
plasma drug concentration of propofol | measured during the perioperative period
  Plasma concentration over time will be measured and modeled in order to calculate drug clearance, volume of distribution, area under the curve, and micro rate constants.
  Knowledge of these variables will allow safer administration of anesthetic drug administration in the obese population. Knowledge of these parameters will allow propofol to be administered safely in morbily obese subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Ingrande, M.D., M.S., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Ingrande J, Gabriel RA, McAuley J, Krasinska K, Chien A, Lemmens HJM. The Performance of an Artificial Neural Network Model in Predicting the Early Distribution Kinetics of Propofol in Morbidly Obese and Lean Subjects. Anesth Analg. 2020 Nov;131(5):1500-1509. doi: 10.1213/ANE.0000000000004897. PMID 33079873